CLINICAL TRIAL: NCT06867224
Title: Transcranial Ultrasound Stimulation as a Neuromodulation Therapy for Craving and Relapse Behaviors in Alcohol Use Disorder.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JDu-014
Record Dates: First submitted 2025-02-20; First posted 2025-03-10 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Use Disorder (AUD); Transcranial Ultrasound Stimulation
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The active group will receive active transcranial ultrasound stimulation.
  Interventions: Device: Active TUS-vmPFC
- Control group (Sham Comparator): The sham group will receive shame transcranial ultrasound stimulation.
  Interventions: Device: Shame TUS-vmPFC

INTERVENTIONS:
Device: Shame TUS-vmPFC — The sham stimulation protocol maintained identical parameter settings to the active treatment group with equivalent application of ultrasound coupling gel at the left vmPFC site localized via the FP1 electrode. Crucially, the ultrasound transducer's output trigger was disabled during sham sessions, ensuring identical device operation procedures without acoustic energy delivery. Participants received daily 15-minute sham sessions matching the active group's 10-day treatment schedule.
  Arms: Control group
Device: Active TUS-vmPFC — Participants in the active stimulation group will receive the transcranial ultrasound stimulation (TUS) targeted the left ventromededial prefrontal cortex (vmPFC), localized via the FP1 electrode position of the International 10-20 EEG system. The TUS will be delivered in the form of pulsed sinusoidal waves, with a fundamental frequency of 0.5 MHz and an intensity of 8 W/cm² (spatial peak pulse average intensity [Isppa]). The pulse duration will be 500 microseconds, and the sonication bursts will consist of 50 tone bursts per session, with a duty cycle of 5%. Each burst (pulse repetition frequency: 100 Hz) was followed by an 8-second inter-burst interval, yielding a total session duration of 15 minutes. Participants underwent one daily session for 10 consecutive days.
  Arms: Intervention group

SUMMARY:
This study aims to evaluate the efficacy of transcranial ultrasound stimulation in reducing cravings and preventing relapse in individuals with alcohol use disorders. Utilizing a double-blind design, participants will be randomly assigned to receive either active accelerated transcranial ultrasound stimulation or a sham treatment.

DETAILED DESCRIPTION:
As a major global public health issue, the core therapeutic goal of alcohol use disorder (AUD) is to reduce alcohol craving and prevent relapse. In recent years, transcranial ultrasound stimulation (TUS) has emerged as a reliable non-invasive neuromodulation technique. Studies have shown that abnormalities in neural activity and structure in the ventromedial prefrontal cortex (vmPFC) of AUD are closely associated with alcohol craving and dysregulation of the reward system. However, existing research on non-invasive neuromodulation techniques for AUD has primarily focused on other brain regions, with limited exploration of interventions targeting the vmPFC. This study aims to evaluate the efficacy of a TUS intervention targeting the vmPFC through a randomized controlled trial, assessing its potential to reduce alcohol craving and prevent relapse, thereby providing a theoretical foundation for clinical translation.

ELIGIBILITY:
Inclusion Criteria:

* Education level of junior high school or above, capable of completing questionnaires and behavioral tests;
* Aged 18-60 years;
* Meet DSM-5 diagnostic criteria for Alcohol Use Disorder;
* No abnormal findings on physical examination;
* Agree to participate in follow-up assessments;
* No contraindications for MRI scanning.

Exclusion criteria:

* Have impaired intelligence (Intelligence Quotient<70);
* Prior tDCS or TMS treatment within the past 3 months;
* Contraindications for TMS therapy (e.g., intracranial metal implants, history of traumatic brain injury, skull defects, cardiac pacemakers, cardiovascular diseases, or epilepsy);
* Severe somatic diseases or major organ dysfunction;
* Psychiatric disorders per DSM-5 criteria (e.g., schizophrenia, schizoaffective disorder, intellectual disability, autism spectrum disorder, dementia, memory impairment, or other cognitive disorders);

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
The change of alcohol craving | baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Alcohol craving was assessed using the Visual Analog Scale (VAS; 0-10 points, higher scores indicating greater craving) during dual-condition olfactory exposure. Participants completed sequential 1.5-minute sniffing trials with alcohol cues and neutral stimuli (water), with the final craving score calculated as the alcohol-induced VAS score minus the neutral-state baseline.
The change of relapse behaviors with alcohol | baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Alcohol consumption and related behaviors were assessed using the Alcohol Use Disorders Identification Test (AUDIT,10 item). Each item is scored from 0 to 4 points, with higher scores indicating greater alcohol consumption.
The change of drinking symptom | baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Drinking symptom will be measured by Obsessive Compulsive Drinking Scale (OCDS), a 14-item scale assessing obsessive and compulsive drinking behaviors. Each item is scored from 0 to 4 points. The total score of OCDS ranged from 0 to 56.

SECONDARY OUTCOMES:
The change of sleep | baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Sleep will be measured by the Pittsburgh Sleep Quality Index (PSQI) rated by both patients and observers. The total score of PSQI ranged from 0 to 21, in which higher scores mean a lower level of sleep quality.
The change of depression | baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  A provider administered questionnaire used to assess remission from depression. The HAMD-17 is a 17-item questionnaire to assess depression severity. Each item is scored from 0-4, with higher scores representing increasing depression severity.
The change of anxiety | baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  The HAMD-14 is a 14-item questionnaire to assess depression severity. Each item is scored from 0-4, with higher scores representing increasing anxiety severity.
The change of self-control | baseline, immediately after the intervention.
  The change of self-control will be measured by the stop-signal task and monetary incentive delay task.

OTHER OUTCOMES:
The Change of Heart Rate Variability | baseline, immediately after the intervention
  Heart rate variability (HRV) was quantified using electrocardiogram (ECG) sensors within a polysomnography.
The Change of Functional Connectivity | baseline, immediately after the intervention
  Resting-state functional magnetic resonance imaging (fMRI) will be used to evaluate changes in functional connectivity between the ventromedial prefrontal cortex (vmPFC) and the nucleus accumbens (NAC), key regions within the brain's reward network. Functional connectivity will be quantified using correlation coefficients between the vmPFC and NAC time series. Data will be aggregated to assess group-level changes in connectivity strength, with a focus on intervention-induced alterations.
The change of EEG | baseline, immediately after the intervention
  Electroencephalography (EEG) data were acquired using a Neuroscan SynAmps2 amplifier and a 64-channel Quick-Cap electrode system. The analysis focused on longitudinal changes in behaviorally-relevant event-related potentials (ERPs) across pre- and post-intervention phases. Specific ERP components (e.g., P300, N200) were measured to assess changes in neural activity associated with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Du, M.D, Ph.D., Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No